CLINICAL TRIAL: NCT03634241
Title: Single-Arm, Phase II of Immunotherapy With Pembrolizumab for the Prevention of Lung Cancer (IMPRINT-Lung)
Brief Title: Pembrolizumab in Preventing Lung Cancer in Patients With Stage I-II Non-Small Cell Lung Cancer or High-Risk Pulmonary Nodules, the IMPRINT-Lung Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-0366; NCI-2018-01588 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0366 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-08-10; First posted 2018-08-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Participants receive pembrolizumab IV over 30 minutes on day 1. Treatment repeat every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scans and collection of blood samples throughout the trial.
  Interventions: Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Procedure: Computed Tomography; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized Axial
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase II trial studies how well pembrolizumab works in preventing lung cancer patients with stage I-II non-small cell lung cancer or high-risk pulmonary nodules. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether immune checkpoint blockade using pembrolizumab eliminates persistent (on two computed tomography [CT] scans at least 3 months apart with no evidence of shrinkage or regression) high-risk indeterminate pulmonary nodules (IPNs) at 6 months after treatment initiation.

SECONDARY OBJECTIVES:

I. To determine whether immune checkpoint blockade using pembrolizumab decreases the incidence of lung cancers confirmed by histology (biopsy or resection).

II. To determine whether immune checkpoint blockade using pembrolizumab prolongs cancer free survival (disease free survival [DFS]) compared with observation in patients with high-risk IPNs.

III. To determine whether immune checkpoint blockade using pembrolizumab prolongs lung cancer-specific survival compared with observation in patients with high-risk IPNs.

IV. To determine whether immune checkpoint blockade using pembrolizumab prolongs overall survival (OS) compared with observation in patients with high-risk IPNs.

V. To assess the safety and tolerability of pembrolizumab in patients with high-risk IPNs.

VI. To assess quality of life patient reported outcomes in patients treated with pembrolizumab compared with patients under observation.

VII. To determine whether immune checkpoint blockade using pembrolizumab decreases the solid component of high-risk IPNs.

VIII. To assess the health-related quality of life (QoL) on subjects enrolled in the study.

EXPLORATORY OBJECTIVES:

I. To explore the radiographic (including radiomic features) evolution of high-risk IPNs with and without treatment of pembrolizumab and to assess their association with risks of risk of lung cancer as well as their association with clinical benefit/toxicities in patients treated with pembrolizumab.

II. To explore the germline deoxyribonucleic acid (DNA) profile and genomic evolution of circulating tumor DNA (ctDNA) of patients with high-risk IPNs and assess their association with risks of risk of lung cancer as well as their association with clinical benefit/toxicities in patients treated with pembrolizumab.

III. To explore the T cell receptor (TCR) repertoire evolution of patients with high-risk IPNs and assess their association with risks of risks of lung cancer as well as their association with clinical benefit/toxicities in patients treated with pembrolizumab.

IV. To explore the evolution of serum soluble factors, such as IFN-gamma and interferon inducible factors (such as CXCL9 and CXCL10), IL-12, TNFalpha, IL-10, TGF-beta, VEGF, IL-6, IL-8, IL-17, IL-18, C-reactive protein etc. and assess their association with risks of risks of lung cancer as well as their association with clinical benefit/toxicities in patients treated with pembrolizumab.

V. To explore the evolution of immunophenotyping or characterization of the immune cell subsets in the periphery, including, but not limited to, T cells, B cells, natural killer [NK] cells, or subpopulations of the aforementioned immune cell types and assess their association with risks of risks of lung cancer as well as their association with clinical benefit/toxicities in patients treated with pembrolizumab.

VI. To explore the evolution of microbiome and assess their association with risks of lung cancer as well as their association with clinical benefit/toxicities in patients treated with pembrolizumab.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeat every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) scans and collection of blood samples throughout the trial.

After conclusion of study treatment, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with no history of lung cancer, who have IPNs detected by LDCT-guided lung cancer screening or imaging studies for other reasons (incidentalomas) with 10 - 30% cancer probability by Brock University cancer prediction equation as following47. This is one of the most frequently utilized cancer risk prediction equations and has been confirmed to be highly effective in catching the disease in its very early stages by large national studies.
2. Participants with no history of lung cancer, who have IPNs detected by LDCT-guided lung cancer screening or imaging studies for other reasons (incidentalomas) with > 30% cancer probability by Brock University cancer prediction equation as following, but biopsy reveals no clear evidence of malignancy.
3. Participants with history of stage I-II non-small cell lung cancer (NSCLC), who have completed curative treatment (surgery and/or radiation) with or without chemotherapy, who have persistent IPNs (on two CT scans at least 3 months apart with no evidence of shrinkage or regression) with 5-30% cancer probability by Brock University cancer prediction equation as following.
4. Participants with history of stage I-II NSCLC, who have completed curative treatment (surgery and/or radiation) with or without chemotherapy, who have persistent IPNs (on two CT scans at least 3 months apart with no evidence of shrinkage or regression) with > 30% cancer probability by Brock University cancer prediction equation as following, but biopsy reveals no clear evidence of malignancy.
5. Persistent IPNs with estimated cancer probability ≥ 5% AND at least one of the following criteria

i. Emergence of solid components within 12 months before the time of screening for patients with pure GGO nodules OR ii. Enlargement of solid components within 12 months before the time of screening for patients with partial solid nodules OR iii. Enlargement of the overall size of lung nodule leading to increase in predicted risk by 5% within 12 months before the time of screening 2. Male/female participants who are at least 18 years of age on the day of signing informed consent with diagnosis of high-risk IPNs as defined below will be enrolled in this study.

3. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 12 weeks while receiving pembrolizumab plus an additional 120 days (a spermatogenesis cycle) for study treatments with evidence of genotoxicity at any dose after the last dose of study treatment and refrain from donating sperm during this period.

4. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days for study treatments with risk of genotoxicity after the last dose of study treatment.

   5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.

   6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of study enrollment.

   7. Have adequate organ function as defined in the following table (Table 4). Specimens must be collected within 10 days prior to the start of study treatment.

   Table 4 Adequate Organ Function Laboratory Values Hematological
   * Absolute neutrophil count (ANC) = ≥1500 per microliter (within 10 days prior to the start of study treatment).
   * Platelets = ≥100,000 per microliter (within 10 days prior to the start of study treatment).
   * Hemoglobin = ≥ 9.0 grams per microliter or = ≥ 5.6 millimoles/liter (within 10 days prior to the start of study treatment) (*criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks).
   * Creatinine OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCL]) =≤ 1.5 x ULN OR = ≥ 30 milliliters per minute (min) for participant with creatinine levels > 1.5 x institutional upper limit of normal (ULN) (creatinine clearance (CrCl) should be calculated per institutional standard.) (within 10 days prior to the start of study treatment).
   * Total bilirubin = ≤ 1.5 x ULN OR direct bilirubin = ≤ ULN for participants with total bilirubin levels > 1.5 x ULN (within 10 days prior to the start of study treatment).
   * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) = ≤ 2.5 x ULN (within 10 days prior to the start of study treatment).
   * International normalized ratio (INR) OR prothrombin time (PT), activated partial thromboplastin time (aPTT) = ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (within 10 days prior to the start of study treatment).

     * PT(INR), aPTT only required for patients having a biopsy and/or if clinically indicated

   Exclusion Criteria:
   * Participant has lung diseases currently requiring oxygen supplement.
   * Participants has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
   * Participant has other lung diseases requiring steroids treatment (10mg of prednisone or equivalent) within 4 weeks at the time of screening.
   * A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
   * Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
   * Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to treatment. Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
   * Has received prior chest radiotherapy and the radiation field overlaps with IPNs. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
   * Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
   * Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
   * Has a known additional metastatic malignancy that is progressing or requiring active treatment. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ), or potentially curable early-stage malignancies including localized NSCLC, head and neck squamous carcinoma, breast cancer, bladder cancer etc., that have undergone potentially curative therapy (surgery and/or radiation with or without chemotherapy) are not excluded.
   * Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
   * Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
   * Has an active infection requiring systemic therapy.
   * Has a known history of Human Immunodeficiency Virus (HIV).
   * Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
   * Has a known history of active TB (Bacillus Tuberculosis).
   * Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
   * Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
   * Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Regression rate of high-risk indeterminate pulmonary nodules (IPNs) | At 6 months
  This will be estimated by the Kaplan-Meier method.

SECONDARY OUTCOMES:
Incidence of lung cancer | Up to 6 months
  This will be estimated by the Kaplan-Meier method.
Cancer-free survival | Up to 6 months
  Stratified log-rank test will be used to compare cancer-free survival between treatment groups. The Cox (proportional hazards) regression model will be used to incorporate potential prognostic factors and treatment assignments as covariates.
Lung cancer-specific survival | Up to 6 months
  Stratified log-rank test will be used to compare cancer-free survival between treatment groups. The Cox (proportional hazards) regression model will be used to incorporate potential prognostic factors and treatment assignments as covariates.
Overall survival | Up to 6 months
Incidence of adverse events | Up to 6 months
  A Bayesian method to monitor the toxicity in the perioperative phase will be used. Toxicity data will be summarized by frequency tables.
Quality of life questionnaires | Up to 6 months
  1. European Organization for Research and Treatment of Cancer Quality of Life of Questionnaire- Cancer 30 (EORTC QLQ-C30).
  2. European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 29 Module ( EORTC QLQ-LC29).
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Zhang, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org